CLINICAL TRIAL: NCT02665065
Title: A Multicenter, Pivotal Phase 3 Study of Iomab-B Prior to Allogeneic Hematopoietic Cell Transplant Versus Conventional Care in Older Subjects With Active, Relapsed or Refractory Acute Myeloid Leukemia (AML)
Brief Title: Study of Iomab-B vs. Conventional Care in Older Subjects With Active, Relapsed or Refractory Acute Myeloid Leukemia
Acronym: SIERRA
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Actinium Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Iomab-01
Record Dates: First submitted 2016-01-22; First posted 2016-01-27 (Estimated); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Acute Myeloid Leukemia; Leukemia, Acute Myeloid; Myeloid Leukemia, Acute; Leukemia, Myeloid, Acute; Acute Myelogenous Leukemia; Leukemia, Acute Myelogenous; Myelogenous Leukemia, Acute; AML; Bone Marrow Transplant
Keywords: Acute Myeloid Leukemia; Leukemia, Acute Myeloid; Myeloid Leukemia, Acute; Bone Marrow Cell Transplant; Transplant, Bone Marrow; HCT; HSCT; Refractory AML; Relapsed AML; BC8; I-131; Iomab; Iomab-B; CD45; Iodine; Iodine-131; 131-I; AML; BMT; Radioimmunotherapy
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Iomab-B (Experimental): Iomab-B in conjunction with a Reduced Intensity Conditioning (RIC) regimen containing Fludarabine and low-dose Total Body Irradiation (TBI) prior to allogeneic HCT
  Interventions: Drug: Iomab-B; Procedure: HCT
- Conventional Care (Active Comparator): Defined as Investigator's choice of salvage chemotherapy with any combination of the following agents: Azacitidine (not allowed as a single agent), Carboplatin, Cladribine, Clofarabine, Cyclophosphamide, Cytarabine, Daunorubicin, Decitabine (not allowed as a single agent with the exception of patients with documented TP53 mutations who have not previously received 10-day regimens of single agent decitabine), Doxorubicin, Enasidenib, Etoposide, Fludarabine, Gemtuzumab ozogamicin, Idarubicin, Ivosidenib (for subjects with IDH1 mutation), L-Asparaginase, Midostaurin (for FLT3 mutant or FLT3-ITD subjects only, not allowed as single agent), Mitoxantrone, Sorafenib (for FLT3 mutant or FLT3-ITD subjects only, not allowed as single agent), Thioguanine, Topotecan, Venetoclax (in combination with a hypomethylating agent). Chemotherapy agents not listed above may be administered after providing clinical justification and receiving medical monitor approval prior to initiation of treatment.
  Interventions: Drug: Conventional Care; Procedure: HCT

INTERVENTIONS:
Drug: Iomab-B
  Arms: Iomab-B
Drug: Conventional Care
  Arms: Conventional Care
Procedure: HCT

SUMMARY:
The primary objective of this study is to demonstrate the efficacy of Iomab-B, in conjunction with a Reduced Intensity Conditioning (RIC) regimen and protocol-specified allogeneic hematopoietic stem cell transplant (HCT), versus Conventional Care in patients with Active, Relapsed or Refractory Acute Myeloid Leukemia (AML).

DETAILED DESCRIPTION:
SIERRA is a pivotal Phase 3 randomized controlled study of Iomab-B in Relapsed or Refractory AML patients. The SIERRA trial has a primary endpoint of durable Complete Remission (dCR) at six months and a secondary endpoint of overall survival following randomization to Iomab-B, as well as Event-Free Survival. Iomab-B is intended to prepare and condition patients for a bone marrow transplant, also referred to as a hematopoietic stem cell transplant, in a potentially safer and more efficacious manner than intensive chemotherapy conditioning that is the current standard of care in bone marrow transplant conditioning.

ELIGIBILITY:
Inclusion Criteria:

* Have active, relapsed or refractory Acute Myeloid Leukemia (AML). Active, relapsed or refractory AML is defined as any one of the following (1) primary induction failure, or (PIF) after 2 or more cycles of therapy, or (2) first early relapse after a remission duration of fewer than 6 months, or (3) relapse refractory to salvage combination chemotherapy, or (4) second or subsequent relapse
* Have documented CD45 expression by leukemic cells via flow cytometry (a "blast gate" on CD45 vs. side scatter analysis consistent with AML)
* Be at least 55 years of age
* Have a circulating blast count of less than 10,000/mm3 (control with hydroxyurea is allowed)
* Have a calculated creatinine clearance (Cockcroft-Gault equation) > 50 mL/min
* Have adequate hepatic function (direct bilirubin, aspartate aminotransferase (AST), and alanine aminotransferase (ALT), defined as ≤ 2 times the upper limit of normal [ULN])
* Have a Karnofsky score ≥ 70
* Have an expected survival of > 60 days
* Have a central venous catheter line in place prior to study treatment administration
* Have 8/8 allele-level, related or unrelated, medically cleared HSC donor matching at human leukocyte antigen (HLA)-A, HLA-B, HLA-C, and DRB-1 with a donor who is medically cleared. Syngeneic donors that meet these criteria are allowed
* Women of childbearing potential, be surgically sterile or agree to practice abstinence or utilize acceptable contraception (intrauterine, injectable, transdermal, or combination oral contraceptive) through 1-year post transplant; Males who are sexually active with women of childbearing potential must be surgically sterile or using an acceptable method of contraception (defined as barrier methods in conjunction with spermicides) from time of screening through 12 weeks after last dose of study drug
* Be able to understand the study procedures, agree to participate in the study program, and voluntarily provide written Informed Consent

Exclusion Criteria:

* Have circulating HAMA noted on initial screening
* Have received prior radiation to maximally tolerated levels to any critical normal organ
* Have active leukemic central nervous system (CNS) involvement, as defined by any leukemic blasts detected in the cerebrospinal fluid (CSF) by morphology or flow cytometry and/or any chloromas detected by CNS imaging
* Have previously received HCT (including both allogeneic and autologous HCT)
* Have clinically significant cardiac disease (NYHA Class III or IV); clinically significant arrhythmia i.e. ventricular tachycardia, ventricular fibrillation, or "Torsade de Pointes". Myocardial infarction with uncontrolled angina within 6 months, congestive heart failure, or clinically significant cardiomyopathy
* Have abnormal QTcF (>450milliseconds) after electrolytes have been corrected (at least two different ECG readings and at least 15 minutes between readings). Subjects with paced rhythm or prolonged QTcF may be exempt from this exclusion if considered eligible for transplant per treating physician clinical judgement with optional cardiology consultation
* Have current or prior positive test results for human immunodeficiency virus (HIV) or hepatitis B (HBV) or C. Subjects who have positive HBV test results due to having been previously vaccinated against hepatitis B, as evidenced by negative hepatitis B surface antigen (HBsAg), negative anti- hepatitis B core protein (HBc) and positive antibody to the HBsAg (anti-HBs) are not excluded. Subjects who have positive hepatitis test results with adequate organ function as defined in the protocol are not excluded
* Have active serious infection uncontrolled by antibiotics or antifungals
* Have acute promyelocytic leukemia and the associated cytogenic translocation t(15/17)
* Have active malignancy within 2 years of entry. Active malignancy is defined as those malignancies requiring treatment with anti-cancer therapy or in the event of indolent malignancies, having measurable disease. Exceptions to this exclusion include: myelodysplastic syndrome, treated non-melanoma skin cancer, completely resected Stage 0 or 1 melanoma no less than 1 year from resection, carcinoma in situ or cervical intraepithelial neoplasia, and successfully treated organ-confined prostate cancer with no evidence of progressive disease based on prostate specific antigen (PSA) levels and are not on active therapy
* Have a perceived inability to tolerate diagnostic or therapeutic procedures, particularly treatment in radiation isolation
* Currently receiving any other active investigational agents

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2016-06; Primary Completion 2022-06 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Durable Complete Remission (dCR) | 6 months from time of initial CR or CRp
  Defined as CR or CRp lasting 180 days or more from time of initial CR or CRp is documented with evidence of subsequent relapse

SECONDARY OUTCOMES:
Overall Survival (OS) following randomization to Iomab-B versus Convetional Care | Over a 5 year period
  Patient overall survival
Event-Free Survival | Over a 5 year period
  Duration of time from randomization to the date of induction treatment failure (ITF), relapse or death

CONTACTS AND LOCATIONS:
Overall Officials: Avinash Desai, MD, Study Chair — Actinium Pharmaceuticals
Locations (24):
- United States (22):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Yale Cancer Center, New Haven, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Mayo Clinic, Jacksonville, Florida
  - Loyola University Medical Center, Maywood, Illinois
  - University of Iowa, Iowa City, Iowa
  - The University of Kansas Cancer Center, Westwood, Kansas
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Roswell Park Cancer Institute, Buffalo, New York
  - Weill Cornell Medicine, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Stony Brook University, Stony Brook, New York
  - University of North Carolina Hospital, Chapel Hill, North Carolina
  - University Hospital of Cleveland Seidman Cancer Center, Cleveland, Ohio
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (2):
  - University of Ottawa, Ottawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario

REFERENCES:
- [Derived] Gyurkocza B, Nath R, Seropian S, Choe H, Litzow MR, Abboud C, Koshy N, Stiff P, Tomlinson B, Abhyankar S, Foran J, Hari P, Chen G, Al-Kadhimi Z, Kebriaei P, Sabloff M, Orozco JJ, Jamieson K, Silverman M, Van Besien K, Schuster M, Law AD, Larkin K, Pandit-Taskar N, Rowley SD, Munshi P, Cook R, Levy MY, Lazarus HM, Sandmaier BM, Pagel JM, Reddy V, MacDougall J, McNamara K, Spross J, Haeuber E, Vusirikala M, Nahar A, Desai A, Giralt S. Randomized Phase III SIERRA Trial of 131I-Apamistamab Before Allogeneic Hematopoietic Cell Transplantation Versus Conventional Care for Relapsed/Refractory AML. J Clin Oncol. 2025 Jan 10;43(2):201-213. doi: 10.1200/JCO.23.02018. Epub 2024 Sep 19. PMID 39298738
- [Derived] Walter RB. Where do we stand with radioimmunotherapy for acute myeloid leukemia? Expert Opin Biol Ther. 2022 May;22(5):555-561. doi: 10.1080/14712598.2022.2060735. Epub 2022 Mar 31. PMID 35350938